CLINICAL TRIAL: NCT01720537
Title: A Phase I, Placebo-Controlled, Randomized Study To Assess The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Following Single, Ascending Doses Of PF-05335810 In Hypercholesterolemic Subjects, With One, Open-Label, Multiple Fixed Dosage Cohort
Brief Title: A Study To Assess The Safety Of PF-05335810 In Hypercholesterolemic Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: B3091001
Record Dates: First submitted 2012-08-03; First posted 2012-11-02 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Hypercholesterolemia
Keywords: High Cholesterol; Dyslipidemia
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias | interventions — bococizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental)
  Interventions: Biological: PF-05335810 Dose A
- Cohort 2 (Experimental)
  Interventions: Biological: PF-05335810 Dose B; Biological: Placebo; Biological: PF-04950615 Dose A
- Cohort 3 (Experimental)
  Interventions: Biological: PF-05335810 Dose C; Biological: Placebo; Biological: PF-04950615
- Cohort 4 (Experimental)
  Interventions: Biological: PF-05335810 Dose D; Biological: Placebo
- Cohort 5 (Experimental)
  Interventions: Biological: PF-05335810 Dose E
- Cohort 6 (Experimental)
  Interventions: Biological: PF-05335810 Dose D; Biological: Placebo

INTERVENTIONS:
Biological: PF-05335810 Dose A — Single SC Injection
  Arms: Cohort 1
Biological: PF-05335810 Dose B — Single Subcutaneous Injection(s)
  Arms: Cohort 2
Biological: Placebo — Single Subcutaneous Injection(s)
  Arms: Cohort 2
Biological: PF-05335810 Dose B — Single Intravenous Infusion
  Arms: Cohort 2
Biological: Placebo — Single Intravenous Infusion
  Arms: Cohort 2
Biological: PF-04950615 Dose A — Single Subcutaneous Injection(s)
  Arms: Cohort 2
Biological: PF-04950615 Dose A — Single Intravenous Infusion
  Arms: Cohort 2
Biological: PF-05335810 Dose C — Single Subcutaneous Injection(s)
  Arms: Cohort 3
Biological: Placebo — Single Subcutaneous Injection(s)
  Arms: Cohort 3
Biological: PF-05335810 Dose C — Single Intravenous Infusion
  Arms: Cohort 3
Biological: Placebo — Single Intravenous Infusion
  Arms: Cohort 3
Biological: PF-04950615 — Single Subcutaneous Injection(s)
  Arms: Cohort 3
Biological: PF-05335810 Dose D — Single Subcutaneous Injection(s)
  Arms: Cohort 4
Biological: Placebo — Single Subcutaneous Injection(s)
  Arms: Cohort 4
Biological: PF-05335810 Dose E — Multiple fixed dosages administered in subcutaneous injections, monthly for 3 months.
  Arms: Cohort 5
Biological: PF-05335810 Dose D — Single Intravenous Infusion
  Arms: Cohort 6
Biological: Placebo — Single Intravenous Infusion
  Arms: Cohort 6

SUMMARY:
This study is to evaluate the safety, tolerability and immunogenicity of single, ascending or multiple fixed subcutaneous and intravenous administrations of PF 05335810 to hypercholesterolemic subjects when added on to a daily statin dose.

ELIGIBILITY:
Inclusion Criteria:

* On stable daily doses of a statin for 45 days prior to receiving study treatment.
* Fasting LDL C equal or greater than 80 mg/dL at screening and visit approximately 1 week prior to randomization.

Exclusion Criteria:

* History of a cardiovascular or cerebrovascular event or procedure within one year of randomization.
* Poorly controlled type 1 or type 2 diabetes mellitus (defined as HbA1c >9%).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2012-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to Day 85/169 or Early Termination (ET)
  Counts of participants who had treatment-emergent adverse events (TEAEs), defined as newly occurring or worsening after first dose. Relatedness to [study drug] was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Number of Participants With Laboratory Test Values of Potential Clinical Importance | Baseline up to Day 85/169 or Early Termination (ET)
  Pre-defined criteria were established for each laboratory test to define the values that would be identified as of potential clinical importance.
Change From Baseline in Heart Rate | Baseline, Day 1 to 85/169 or ET
Diastolic Blood Pressure | Baseline, Day 1 to 85/169 or ET
Change From Baseline in Electrocardiogram (ECG) Parameters | Baseline, Day 1 to 85/169 or ET
Number of Participants With Laboratory Test Values of Potential Clinical Importance | Baseline, Day 1 to 85/169 or ET
  Pre-defined criteria were established for each laboratory test to define the values that would be identified as of potential clinical importance.

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | Day1 pre-dose to Day 85/169 or ET
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] | Day1 pre-dose to Day 85/169 or ET
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)
Maximum Observed Plasma Concentration (Cmax) | Day1 pre-dose to Day 85/169 or ET
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Day1 pre-dose to Day 85/169 or ET
Apparent Volume of Distribution (Vz/F) | Day1 pre-dose to Day 85/169 or ET
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Apparent Oral Clearance (CL/F) | Day1 pre-dose to Day 85/169 or ET
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Plasma Decay Half-Life (t1/2) | Day1 pre-dose to Day 85/169 or ET
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Absolute Bioavailability (%F) | Day1 pre-dose to Day 85/169 or ET

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (7):
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, San Antonio, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3091001&StudyName=A%20Study%20To%20Assess%20The%20Safety%20Of%20PF-05335810%20In%20Hypercholesterolemic%20Subjects